CLINICAL TRIAL: NCT03756493
Title: The Added Benefit of L-PRF to Autogenous Bone Graft in the Treatment of Degree II Furcation Involvements in Mandibular Molars
Brief Title: Added Benefit of L-PRF to Autogenous Bone Graft in the Treatment of Mandibular Degree II Furcation Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, full time professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11042017
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Periodontal Attachment Loss; Periodontal Bone Loss
Keywords: Platlet rich fibrin; Bone graft; Furcation defects
MeSH Terms: conditions — Periodontal Attachment Loss; Alveolar Bone Loss; Furcation Defects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OFD+ABG+L-PRF treated patients (Experimental): Periodontal surgery with Leukocyte and Platelet Rich Fibrin (L-PRF) is performed, after local anaesthesia, mucoperiosteal SPPFs will be raised. Autogenous bone graft mixed with cutted L-PRF will be applied to the furcation defects; then, a L-PRF membrane is positioned above the filling material. Finally the flap will be coronally positionated and sutured by interrupted sutures.
  Interventions: Procedure: Periodontal Surgery with OFD+ABG+L-PRF
- OFD+ABG treated patients (Active Comparator): Periodontal surgery with Autogenous Bone Graft (ABG) is performed, after local anaesthesia, mucoperiosteal SPPFs will be raised. ABG will be applied to the furcation defects. Finally the flap will be coronally positioned and sutured by interrupted sutures.
  Interventions: Procedure: Periodontal Surgery with OFD+ABG
- OFD treated patients (Active Comparator): Periodontal surgery with Open Flap Debridement is performed, after local anaesthesia, mucoperiosteal SPPFs will be raised. No grafts will be applied to the furcation defects. Finally the flap will be coronally positioned and sutured by interrupted sutures.
  Interventions: Procedure: Periodontal Surgery OFD

INTERVENTIONS:
Procedure: Periodontal Surgery with OFD+ABG+L-PRF — Patients will be treated by periodontal surgical flaps with the addition of L-PRF+ Autogenous Bone Graft filling material.
  Arms: OFD+ABG+L-PRF treated patients
Procedure: Periodontal Surgery with OFD+ABG — Patients will be treated by periodontal surgical flaps with the addition of Autogenous Bone Graft filling material.
  Arms: OFD+ABG treated patients
Procedure: Periodontal Surgery OFD — Patients will be treated by Open Flap Debridement without use of filling material.
  Arms: OFD treated patients

SUMMARY:
Different therapeutic approaches have been proposed for the treatment of furcation defects and the regeneration of periodontium within the furcation area is considered one of the most challenging aspect of surgical periodontal therapy.

Periodontal regeneration is a highly predictable therapeutic option for the treatment of different furcation defects, particularly class II furcation involvements in the lower molars.

In particular, the application of a combined therapeutic approach (i.e., barrier, bone re-placement graft with or without biological agents) seems to offer better results as compared with monotherapeutic treatments.

Several studies have demonstrated that platelet concentrates, such as platelet-rich plasma (PRP), platelet-derived growth factor (PDGF) and, more recently, leukocyte and platelet-rich fibrin (L-PRF) can represent new therapeutic options for bone regeneration procedures by increasing the healing potential of natural blood clot in the surgical site.

Leukocyte and Platelet-rich fibrin (L-PRF) is a second-generation platelet concentrate, developed by Choukroun et al. It is prepared without the addition of any anticoagulants and consists of a slowly polymerized complex fibrin network which incorporates leukocytes, glycan chains, structural glycoproteins and an high concentration of growth factors such as transforming growth factor β (TGF-B), platelet-derived growth factor (PDGF), vascular endothelial growth factor (VEGF). The three-dimensional architecture and the specific biochemical properties, which facilitate the wound healing processes, have led to a widespread use of this biomaterial in plastic surgery, maxillofacial surgery, oral and periodontal surgery.

A large clinical and histological evidence supports the concept that autogenous bone grafts (ABG) are highly effective regenerative materials in the treatment of intrabony defects. Moreover, with respect to the treatment of furcation defects, outcome data from a number of studies generally indicate positive clinical benefits with the use of bone grafts in the treatment of Class II furcations.

Therefore, on the basis of such considerations, the aim of this study was to evaluate the effectiveness of a combined regenerative treatment by L- PRF and ABG in the treatment of mandibular molars degree II furcation defects and to compare the outcomes of such a treatment with those from (OFD)+ABG and OFD alone treatments.

DETAILED DESCRIPTION:
Experimental Design. This randomized, comparative and clinical trial will be designed to evaluate the clinical and radiographic outcomes 6 months after three treatment modalities of mandibular degree II furcation defects.

The patients study will exhibit buccal or lingual mandibular degree II furcation defects; all experimental sites will be accessed with a SPPF procedure. L- PRF and autogenous bone graft (ABG) will be applied to the debrided defects in the OFD+ABG+L-PRF group; the OFD+ABG group will receive only ABG and the OFD group will be treated with Open Flap Debridement (OFD) alone.

Study Population. At least fifty-four patients, aged 18 to 70 years old, affected by moderate-to-severe chronic periodontitis, will be selected for this study and treated at the Operating Unit of Periodontology and Oral Hygiene of the Department of Medical, Oral and Biotechnological Sciences, "G. D'Annunzio" Chieti-Pescara University, Italy. Each patient will participate in the study with a single experimental site.

The participants will receive verbal and written information and will sign a consent form approved by the Ethical Committee of the G. D'Annunzio University of Chieti medical faculty. The study protocol is in accordance with the Declaration of Helsinki of 1975, as revised in 2013.

Each defect will be assigned a defect number and will be randomly allocated to one of the three treatment regimens. Assignment will be performed by a custom made computer-generated table. To conceal allocation, opaque envelops will be assigned to the specific experimental site and will be opened during surgery.

Four months before the surgical treatment, all 54 patients will undergo non-surgical periodontal treatment consisting of supragingival and subgingival scaling and root planing (SRP) by ultrasonic instruments and hand curets and motivational instructions on oral home care.

Complete oral and periodontal examinations will be performed for each patient before and 4 months after the non-surgical treatment. These will include full mouth plaque score (FMPS), full mouth bleeding score (FMBS), probing depth (PD), vertical clinical attachment level (VCAL), horizontal clinical attachment level (HCAL), and gingival recession (GR) for six sites per tooth (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual/ palatal, mid-lingual/palatal, and disto-lingual/palatal sites). The measurements will be recorded using a University of North Carolina (UNC-15, HuFriedy, Chicago, Illinois, USA) periodontal probe.

Clinical measurements at mid-buccal or mid-lingual experimental sites will be taken immediately before surgical treatment (baseline) and 6 months after treatment, by the same experienced examiner (MP), who will be masked to the treatment. The primary outcome of the study will be HCAL gain at 6 months.

Radiographic Measurements. Preoperative and 6 months postoperative standardized radiographs will be taken by the paralleling technique using an individual film-holder device consisting of a bite block rigidly connected to an acrylic dental splint to achieve identical film placement at each evaluation.

The radiographs will be digitized using an image processing device, after choosing the standard scan settings (600 dots per inch and 256 levels of gray).

Measurements related to vertical bone level (VBL) will be performed using a dedicated software and calculating the distance between the furcation fornix and the bottom of the defect.

Before surgery, from each patient of all groups, to avoid unblinding, 30 ml of blood was collected in three 10-ml sterile tubes without anticoagulant, and it was quickly centrifuged‖‖ at 3,000 revolutions/minute for 10 minutes.The fibrin clot (L-PRF) was collected and squeezed in the L-PRF Box to form three membranes.

Surgical Technique. All the surgeries will be performed by the same experienced clinician. In all groups, after local anaesthesia, mucoperiosteal SPPFs will be raised. Mesial and distal vertical releasing incisions will be performed to allow more visibility and defects accessibility. After flap elevation, flap mobility will be tested to ensure that primary closure of the wound could be achieved through tension-free suturing. The granulation tissue adherent to the alveolar bone will be removed to provide full access and visibility to the root and bone surfaces. SRP will be performed. ABG material will be collected using bone scrapers in OFD+ABG+L-PRF group and OFD+ABG group.

In the OFD+ABG+L-PRF group , one L-PRF membrane cutted into small pieces and mixed with ABG will be placed in the furcation defect. The other PRF membranes in each patient will be placed over the grafted defect and will be sutured with an absorbable suture. The OFD+ABG group defects will be grafted only with ABG and will be not covered by a L-PRF membrane. The OFD group defect will be treated only with open flap debridement. Finally the flap will be repositioned and horizontal mattress and interrupted sutures will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* a Full-Mouth Plaque Score (FMPS) and a Full-Mouth Bleeding Score (FMBS) < 20% at the time of surgery;
* to have at least 20 teeth;
* at least 1 mandibular molar with buccal or lingual degree II furcation defects, with no mobility and with horizontal CAL (HCAL) > 3 mm and vertical probing depth in the central-vestibular or central-lingual site >= 5 mm after non surgical treatment.

Exclusion Criteria:

* systemic diseases;
* medications affecting periodontal status during the previous 6 months;
* pregnant or lactating;
* smokers;
* periodontal therapy in the 2 previous years;
* periapical endodontic lesions;
* dental mobility.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Horizontal Clinical Attachment Gain | 6 months
  The periodontal probe was inserted into the furcation area, perpendicular to a horizontal one which was placed on the buccal or lingual aspect of the involved tooth.

SECONDARY OUTCOMES:
Vertical Bone Level | 6 months
  Radiographic distance between the fornix of furcation and the bottom of the defect.
Vertical Clinical Attachment Gain | 6 months
  Change of the distance between the cementum-enamel junction and the depth of the probable site.
Pocket Probing Depth | 6 months
  Change of the distance between the gingival margin and the depth of the probable site.
Gingival recession | 6 months
  Change of the distance between the cementum-enamel junction and the gingival margin of the probable site.

CONTACTS AND LOCATIONS:
Locations (1):
- G. d'Annunzio University, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: Undecided